CLINICAL TRIAL: NCT01101087
Title: Efficacity of Taurolock in Preventing Primary Bacterial Peritonitis in Patients Undergoing Peritoneal Dialysis for Renal Insufficiency: a Randomized, Multicenter, Double Blind Study With Placebo
Brief Title: Taurolock for Preventing Bacterial Peritonitis During Renal Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PHRC-N/2009/BB; 2009-A00599-48 (Other: RCB number)
Record Dates: First submitted 2010-04-08; First posted 2010-04-09 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Peritonitis; Catheter-related Infections; Renal Insufficiency
Keywords: Dialysis
MeSH Terms: conditions — Peritonitis; Catheter-Related Infections; Renal Insufficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Taurolock (Experimental)
  Interventions: Device: Taurolock
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Taurolock
  Arms: Taurolock
Other: Placebo — Injectable sodium chloride conditioned in exactly the same manner as the experimental product.
  Arms: Placebo

SUMMARY:
Dialysis catheters are sites of bacterial proliferation. The purpose of this study is to determine whether or not the use of Taurolock (a catheter lock solution) can prevent bacterial peritonitis in patients undergoing peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Renal insufficiency, stage V (HAS 2007 classification)
* Requires incident peritoneal dialysis
* No signs of peritoneal infection on inclusion
* signed consent
* affiliated with a social security system

Exclusion Criteria:

* Patient will have a renal transplant in the upcoming year following dialysis
* Survival prognosis for one year is weak
* allergy to citrate, (cyclo)-taurolidine, or heparin
* patient is taking medication with a known contra-indication with citrate or (cyclo)-taurolidine
* patient has a thrombopenia caused by heparin
* impossible to inform the patient correctly
* patient under guardianship
* patient already included in another biomedical research protocol
* no signed consent
* no social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Occurence of bacterial peritonitis | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Branger, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (15):
- France (14):
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, Gard
  - CH d'Avignon - Centre Hospitalier Henri Duffaut, Avignon
  - CHU de Caen - Hôpital Clemenceau, Caen
  - CH de Chambéry, Chambéry
  - CH de Colmar - Hôpitaux Civils de Colmar, Colmar
  - Association CALYDIAL Vienne, Irigny
  - Centre Hospitalier Départemental Vendée - Site de la Roche sur Yon, La Roche-sur-Yon
  - AIDER - Clinque Jacques Mirouze, Montpellier
  - APHP - Groupe Hospitalier Pitié-Salpetrière, Paris
  - CH Pontoise - Centre Hospitalier René Dubos, Pontoise
  - Association AUB Santé Quimper, Quimper
  - Centre Hospitalier Regional - Site Groupe Hospitalier Sud Réunion (GHSR), Saint-Pierre
  - CH de Valenciennes - Hôpital Jean Bernard et Hôtel Dieu, Valenciennes
  - ALTIR - Hôpital Brabois, Vandœuvre-lès-Nancy
- Association APURAD, Paéa, French Polynesia